CLINICAL TRIAL: NCT06491069
Title: Depression, Anxiety and Eating Disorder After Bariatric Surgery
Brief Title: Risk Factors of Depression, Anxiety and Eating Disorder After Bariatric Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Sayed Ali, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-24-05-01MS
Record Dates: First submitted 2024-06-14; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety; Eating Disorders; Bariatric Surgery
MeSH Terms: conditions — Depression; Anxiety Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the goal of this observational study is to Investigate and determine rate of occurrence and associated risk factors of depression , anxiety , eating disorder after bariatric surgery.

participants will undergo psychometric tests.

DETAILED DESCRIPTION:
the aim of this study is to Investigate and determine rate of occurrence and associated risk factors of depression , anxiety , eating disorder after bariatric surgery .

and its correlation to postoperative changes in weight .

All data from the subjects will be obtained through direct interviews of postoperative patients

All subjects will be submitted to :

1. Obtaining detailed history of

Age , sex , socioeconomic level , work , educational level , marital status , functionality of the patient , special habits (smoking index , alchohol and substance abuse , feeding habits , exercise ).

Evaluating the family history of obesity , psychiatric disorder , Bariatric surgery

Searching for early and late complications of Bariatric surgery : Dumping syndrome , malnutrition , vomiting , hernias , redundant ght loss (by wieght skin , skin infection , vomiting .

Determining the type of surgery. degree of obesity of postoperative patients

evaluated by body mass index

Medical comorbidities Hypertension , diabetes , chronic kidney disease , chronic liver disease , ischemic heart disease , obstructive sleep apnea , gastric reflux , dermatological disorders

Psychometric evaluation

Hamilton Anxiety Rating Scale

Hamilton Depression Rating Scale

Eating disorder evaluation. Eating Attitudes Test-26

ELIGIBILITY:
Inclusion Criteria:

* study sample of humans who had bariatric surgery.
* Subjects with postoperative time of ≥ 3 months
* Male or female aged between 18:60 years.

Exclusion Criteria:

* Illiterate patients.
* Patients have dementia or psychosis.
* Age below 18 or above 60 years.
* Patients refused to give written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: the group being investigated is patients who had obesity and underwent Bariatric surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
risk factors of depression , anxiety and rating disorder after bariatric surgery | baseline
  identification of risk factors that lead to occurrence of depression and anxiety and eating disorders in patients who had bariatric surgeris

IPD SHARING:
Plan to Share IPD: Undecided
still undecided

REFERENCES:
- [Background] Sarwer DB, Allison KC, Wadden TA, Ashare R, Spitzer JC, McCuen-Wurst C, LaGrotte C, Williams NN, Edwards M, Tewksbury C, Wu J. Psychopathology, disordered eating, and impulsivity as predictors of outcomes of bariatric surgery. Surg Obes Relat Dis. 2019 Apr;15(4):650-655. doi: 10.1016/j.soard.2019.01.029. Epub 2019 Feb 23. PMID 30858009
- [Background] Brown RM, Guerrero-Hreins E, Brown WA, le Roux CW, Sumithran P. Potential gut-brain mechanisms behind adverse mental health outcomes of bariatric surgery. Nat Rev Endocrinol. 2021 Sep;17(9):549-559. doi: 10.1038/s41574-021-00520-2. Epub 2021 Jul 14. PMID 34262156
- [Background] Ivezaj V, Kessler EE, Lydecker JA, Barnes RD, White MA, Grilo CM. Loss-of-control eating following sleeve gastrectomy surgery. Surg Obes Relat Dis. 2017 Mar;13(3):392-398. doi: 10.1016/j.soard.2016.09.028. Epub 2016 Oct 1. PMID 27913121
- [Background] undefined
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363